CLINICAL TRIAL: NCT01916239
Title: Phase I-II Study of Pomegranate Extract Formulations in Colorectal Cancer Patients: Metabolic and Gene Expression Profiling in Tumoral and Normal Colon Tissues
Brief Title: Pomegranate Extract Supplementation in Colorectal Cancer Patients
Acronym: POMEcolon
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Juan Carlos Espín de Gea, Full Research Professor, National Research Council, Spain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBAS-CSIC-2
Record Dates: First submitted 2013-07-30; First posted 2013-08-05 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Colorectal Cancer
Keywords: Pomegranate; Urolithins; Colorectal cancer; Colon cancer; Metabolite; Gene expression; microRNA; Nutraceutical; Food supplement; Polyphenol; Gut microbiota
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard pomegranate extract formulation (Experimental): Standard pomegranate extract formulation containing 20% punicalagin
  Interventions: Dietary Supplement: Standard pomegranate extract formulation
- Pomegranate extract formulation-1 (Experimental): New pomegranate extract formulation-1
  Interventions: Dietary Supplement: Pomegranate extract formulation-1
- Pomegranate extract formulation-2 (Experimental): New pomegranate extract formulation-2
  Interventions: Dietary Supplement: Pomegranate extract formulation-2

INTERVENTIONS:
Dietary Supplement: Standard pomegranate extract formulation — Standard pomegranate extract formulation containing 20% punicalagin
  Arms: Standard pomegranate extract formulation
Dietary Supplement: Pomegranate extract formulation-1 — New pomegranate extract formulation-1
  Arms: Pomegranate extract formulation-1
Dietary Supplement: Pomegranate extract formulation-2 — New pomegranate extract formulation-2
  Arms: Pomegranate extract formulation-2

SUMMARY:
The most relevant pomegranate phenolics (ellagitannins and ellagic acid) are extensively metabolized by the human gut microbiota to yield a number of metabolites called urolithins (mainly Uro-A). Urolithins have been reported to regulate in vivo the expression of genes involved in inflammation and cancer. Our hypothesis is that urolithins can be detected in the human colon mucosa where these metabolites can exert anti-inflammatory and anti-cancer activities. After colonoscopy and diagnosis, colorectal cancer patients will consume capsules containing three different pomegranate extract formulations until surgery. The aims of this trial are:

* To evaluate the disposition of pomegranate phenolics and urolithins in tumoral and normal colon tissues.
* To evaluate gene expression profiling and protein markers in tumoral and normal colon tissues from these patients.
* To compare different pomegranate extract formulations on the above.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer diagnosis.
* Surgery required.
* WHO status: between 0 and 2.
* Hemoglobin >10 g/dL
* ALT >2.5-fold above the normal value.
* Serum Bilirubin >1.5-fold above the normal value.
* Creatinine <140 micromol/L

Exclusion Criteria:

* Patients who do not satisfy inclusion criteria and,
* Active pectic ulcer.
* Pregnancy or breastfeeding.
* Alcoholism.
* Chemotherapy or radiotherapy a month prior to recruitment.
* Treatment with steroids or other anti-inflammatory drugs a week prior to recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Phenolics and derived metabolites in colon tissues, plasma and urine. | Change from baseline at 15 days
  Occurrence of phenolics and gut-microbiota derived metabolites in tumoral and colon tissues, urine and plasma.
Gene expression profiling in colon tissues | Change from baseline at 15 days
  Gene expression profile changes in tumoral and normal colon tissues

SECONDARY OUTCOMES:
IGF-1 (insulin-like growth factor-1) | Change from baseline at 15 days
  Change in circulating IGF-1 levels
CEA (carcnoembryonic antigen) | Change from baseline at 15 days
  Change in circulating CEA levels
Number of patients with adverse events as a measure of safety and tolerability | Change from baseline at 15 days
  * Change in markers involved in hepatic and renal functions: GGT, AST, ALP, ALT, CPK, urate, creatinin, albumin, bilirubin, LDH.
  * Change in hematological variables: leucocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils, hemoglobin, hematocrit, mean corpuscular volume, mean platelet volume, platelets, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration.
  * Intolerance, dyspepsia, allergic reactions, constipation, diarrhea, abdominal pain, nausea.
microRNA expression profiling in colon tissues | Change from baseline at 15 days
  microRNA (miR) expression profile change in tumoral and normal colon tissues

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Juan Carlos Espín, PhD, Principal Investigator — National Research Council (CEBAS-CSIC, Murcia, Spain)
Locations (1):
- Hospital General Universitario Reina Sofía, Murcia, Murcia, Spain

REFERENCES:
- [Derived] Selma MV, Gonzalez-Sarrias A, Salas-Salvado J, Andres-Lacueva C, Alasalvar C, Orem A, Tomas-Barberan FA, Espin JC. The gut microbiota metabolism of pomegranate or walnut ellagitannins yields two urolithin-metabotypes that correlate with cardiometabolic risk biomarkers: Comparison between normoweight, overweight-obesity and metabolic syndrome. Clin Nutr. 2018 Jun;37(3):897-905. doi: 10.1016/j.clnu.2017.03.012. Epub 2017 Mar 16. PMID 28347564
- [Derived] Nunez-Sanchez MA, Gonzalez-Sarrias A, Garcia-Villalba R, Monedero-Saiz T, Garcia-Talavera NV, Gomez-Sanchez MB, Sanchez-Alvarez C, Garcia-Albert AM, Rodriguez-Gil FJ, Ruiz-Marin M, Pastor-Quirante FA, Martinez-Diaz F, Tomas-Barberan FA, Espin JC, Garcia-Conesa MT. Gene expression changes in colon tissues from colorectal cancer patients following the intake of an ellagitannin-containing pomegranate extract: a randomized clinical trial. J Nutr Biochem. 2017 Apr;42:126-133. doi: 10.1016/j.jnutbio.2017.01.014. Epub 2017 Jan 27. PMID 28183047